CLINICAL TRIAL: NCT04468516
Title: Treatment of Chronic Back Pain With Focused Vibroacoustic Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wilfrid Laurier University (Other)
Collaborators: KKT International (Unknown)
Responsible Party: Principal Investigator, Abdullah Mosabbir, Principal Site Investigator, Wilfrid Laurier University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10010563
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There are two groups (treatment and placebo). Participants will not know which group they are in until the end. Masking will be maintained by the following plan:
  1. Researcher assigning participants to treatment and control groups: Dr. Abdullah Mosabbir.
  2. Researcher(s)/clinician(s) performing pre-treatment/post-treatment assessments: Dr. Aslam Khan, or a Clinician hired by KKT who is NOT doing #3.
  3. Researcher(s)/clinician(s) performing treatments or sham procedure: Dr. Peter Dyback, or a Clinician hired by KKT who is NOT doing #2.
  4. Researcher who will assemble these data, code it, and do the data analysis: Dr. Abdullah Mosabbir.
  5. Researchers who will supervise the design and ethical conduct of the study as well as data analysis: Dr. Heidi Ahonen and Dr. Quincy Almeida.
  6. Researchers whose role is conceptual: Dr.Karim Bayanzay, Dr. Lidan You, and Dr. Lee Bartel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Treatment (Experimental): Intervention is applied to the C1 of the spine.
  Interventions: Device: KKT
- Placebo (Placebo Comparator): Intervention is applied in reduced intensity to the trapezius muscle.
  Interventions: Device: sham KKT
- Waitlist period (No Intervention): Participants will have a 1 month waitlist period where no intervention takes place.

INTERVENTIONS:
Device: KKT — Vibroacoustic sound waves applied focally.
  Arms: Treatment
Device: sham KKT — sham KKT
  Arms: Placebo

SUMMARY:
Chronic back and neck pain is the most common chronic condition worldwide. Unfortunately, the current available treatment options are limited and largely unsuccessful, which is considered as one of the primary drivers for the high cost of back pain management. Systematic reviews show that the results of common treatments including pain medications, surgery, exercise and psychological therapies for back pain demonstrate inconsistent results and moderate improvement. Therefore, non-invasive adjunct therapies can be a useful addition to traditional back pain management.

Focused vibroacoustic treatment for back and neck pain is a non-invasive procedure that applies low frequency sound waves to the spine (50Hz-110Hz), and has shown consistent and positive results in early clinical and animal studies. The goal of this project is to test vibroacoustic sound waves delivered to the spine in a double blind randomized controlled trial to demonstrate the efficacy of focused vibroacoustics in treating chronic back pain.

Participants with back pain will be recruited and divided into a treatment and placebo group and will undergo treatment at a clinic over a one month period. Outcome measures will be collected before and after the intervention period. Placebo participants will be offered the full treatment without charge after the experiment is over.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic low back pain with a disease duration of more than 3 months (further diagnostic results were not required)
* Aged 18-75.
* Scored at least 4/10 in pain scale (VAS or Numerical)
* Written consent

Exclusion Criteria:

* Acute back pain (< 4 weeks)
* History of spinal or vertebral surgery
* History of any vertebral or spinal infection
* History of significant trauma related to the spine
* History of IV drug use
* History of malignancy
* Congenital deformation of the spine (except mild scoliosis or kyphosis)
* Pregnancy
* Previous KKT Treatment
* Undergoing concurrent treatment Unable to complete all 12 treatment sessions due to travel, distance or transportation issues, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of Visual Analog Scale for Pain | 1 month
  A scale which measures the intensity of pain. Scored from 0 to 100. 0 means no pain, 100 means maximum pain.
Change from baseline of Roland Morris Disability Questionnaire | 1 month
  Measures back pain disability.
Change in baseline of EuroQol (EQ5D-5L) Questionnaire | 1 month
  Quality of Life Questionnaire
Change in Neck Pain Disability Index | 1 month
  Measures neck pain disability

SECONDARY OUTCOMES:
Change in Medication Dosage | 1 month
  The assessor will ask what medications the participant is taking. They will record the drug and dosage.
Change in Shoulder and Pelvis tilt | 1 month
  Measured via calipers
Change in Leg length | 1 month
Change in Cervical range of motion | 1 month
Change in Palpatory tenderness of the spine | 1 month
  The assessor will count and record the number of tender regions along the spine.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desmoulin GT, Yasin NI, Chen DW. Spinal mechanisms of pain control. Clin J Pain. 2007 Sep;23(7):576-85. doi: 10.1097/AJP.0b013e3180e00eb8. PMID 17710007
- [Background] Desmoulin GT, Hewitt CR, Hunter CJ. Disc strain and resulting positive mRNA expression from application of a noninvasive treatment. Spine (Phila Pa 1976). 2011 Jun 15;36(14):E921-8. doi: 10.1097/BRS.0b013e3181fd78b3. PMID 21289569
- [Background] Desmoulin GT, Reno CR, Hunter CJ. Free axial vibrations at 0 to 200 Hz positively affect extracellular matrix messenger ribonucleic acid expression in bovine nucleus pulposi. Spine (Phila Pa 1976). 2010 Jul 1;35(15):1437-44. doi: 10.1097/BRS.0b013e3181c2a8ec. PMID 20386503